CLINICAL TRIAL: NCT04566562
Title: Blood Brain Barrier Dysfunction and Postoperative Neurocognitive Disorders in Older Adults
Brief Title: Blood Brain Barrier Dysfunction and Postoperative Neurocognitive Disorders
Acronym: BBBSx
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Rajesh Kumar, PhD, Professor In-Residence, University of California, Los Angeles
Other Study IDs: BBBSx 20-001456
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-08

CONDITIONS: Neurocognitive Disorders; Postoperative Cognitive Dysfunction
Keywords: brain imaging, neurocognitive testing
MeSH Terms: conditions — Neurocognitive Disorders; Postoperative Cognitive Complications | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Brain scans, cognitive tests, blood biomarkers
  Interventions: Diagnostic Test: Brain Imaging; Diagnostic Test: Cognitive Testing; Diagnostic Test: Blood Biomarkers

INTERVENTIONS:
Diagnostic Test: Brain Imaging — Magnetic Resonance Imaging (MRI) using diffusion weighted pseudo-continuous arterial spin labeling (DW-pCASL) .
Diagnostic Test: Cognitive Testing — Wide Range Assessment of Memory and Learning (WRAML 2) and Montreal Cognitive Assessment (MoCA)
Diagnostic Test: Blood Biomarkers — Inflammatory Markers

SUMMARY:
Postoperative neurocognitive disorders (PND), which include postoperative delirium and both acute and longlasting neurocognitive deficits, are a significant public health problem, leading to a cascade of deleterious complications. Older adults are particularly at-risk of developing PND both in the short and long term. Although age is consistently reported as an important risk factor, the exact pathophysiology of PND remains poorly understood, but may include postsurgery-compromised blood brain barrier (BBB) function. This project proposes that perioperative BBB dysfunction is associated with measurable brain morphologic findings in cognitive control areas that can be discovered with non-invasive magnetic resonance imaging (MRI). Patients scheduled for surgery with an age range of 65-75 years of age, will participate in brain diffusion-weighted pseudo-continuous arterial spin labeling (DW-pCASL) and diffusion tensor imaging (DTI), cognitive assessments, and evaluation of a BBB marker from blood (at baseline, at two weeks, and at six months after surgery).

All patients will have a brain scan (MRI) within before surgery and two weeks and six months after surgery. During this visit cognitive function will be assessed. Patients will also be asked to participate in a blood draw.

DETAILED DESCRIPTION:
The investigators will examine the potential mechanisms contributing to PND in an older surgical population. It is proposed that BBB will be altered contributing to brain tissue changes in cognitive control areas that can be examined with MD measures and blood biomarkers. Therefore, the specific aims are to:

AIM #1: Examine BBB function, using DW-pCASL procedures, and BBB marker (S100β levels), in older adult subjects between pre- ) and post-surgery

AIM #2: Assess brain tissue changes, using DTI-based MD measures, and cognition function, between pre- and post-surgery in older adult subjects.

AIM #3: Examine the relationships between BBB blood biomarker, BBB function index, and MD values from cognitive control areas (prefrontal cortex, caudate, and hippocampus) between pre- and post-surgery in an older surgical population.

A One-group comparative and longitudinal study design will be used in this proposal. A total of 34 older subjects scheduled for surgery will be recruited. Patients of either sex, in the age range 65-75 years scheduled for abdominal, gynecologic or urologic.

To assess cognitive function, the WRAML2 and MoCA tests will be performed within one week before surgery and at two weeks and six months after surgery. These tests have been used by our team in several conditions, and will be introduced just before MRI procedures. An average mean score of 100±15 on WRAML2 and a score ≥26 on MoCA will be considered normal.

Examination of BBB integrity from blood. To account for interindividual variation, baseline systemic biomarkers will be measured preoperatively (within one week before surgery). Postoperative samples will also be collected at two weeks and 6 months of surgery. Samples will be batch analyzed using Enzyme-linked immunosorbent assay (S100β) by the UCLA Department of Pathology & Laboratory Medicine.

Magnetic Resonance Imaging. All brain MRI studies will be performed on a 3.0-Tesla MRI scanner (Siemens, Magnetom, Prisma) at the Department of Radiology, UCLA. MRI studies will be performed within one week before surgery, and at two weeks and six months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 65-75 years old
* Scheduled for abdominal, gynecologic or urological surgery

Exclusion Criteria:

* Subjects undergoing surgery with a previous history of stroke, myocardial infarction, current pregnancy (if female), diagnosed neuropsychological and neuropsychiatric diseases, airway or chest deformities that would interfere with breathing, chronic obstructive pulmonary disease, cystic fibrosis, presence of space-occupying brain lesions, any history of drug abuse (e.g., cocaine or tobacco use), chronic kidney disease requiring dialysis.
* Body weight >300 pounds (restrictions of MRI scanner table).
* All subjects with any contraindication to the MRI procedures, such as metallic and electronic implants (phrenic or cardiac pacemakers), claustrophobia, metallic-based tattoos, will also be excluded. Non-english speaking patients will also be excluded as the cognitive tests have not been validated in other languages.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients of either sex, in the age range 65-75 years scheduled for abdominal, gynecologic or urologic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Preoperative cognitive function | pre-surgery (within five days before)
  Montreal Cognitive Assessment (MoCA) test
Postoperative cognitive dysfunction - delayed cognitive recovery | Post-surgery (within two weeks post surgery)
  Montreal Cognitive Assessment (MoCA) test
Postoperative cognitive dysfunction - neurocognitive disorder | Post-surgery (6 months after surgery)
  Montreal Cognitive Assessment (MoCA) test
Preoperative cognitive function II | Pre-surgery (within five days before surgery)
  Wide Range Assessment of Memory and Learning (WRAML2)
Postoperative cognitive dysfunction - delayed cognitive recovery II | Post-surgery (within two weeks post surgery)
  Wide Range Assessment of Memory and Learning (WRAML2)
Postoperative cognitive dysfunction - neurocognitive disorder II | Post-surgery (6 months after surgery)
  Assessment of Memory and Learning (WRAML2)

SECONDARY OUTCOMES:
Blood Serum anti-inflammatory Biomarkers | pre- (within five days before surgery)
  Assess blood inflammatory biomarkers (IL6, TNFa and IL1B) using enzyme-linked immunosorbent assay
Blood Serum anti-inflammatory Biomarkers II | post-surgery (within two weeks of surgery)
  Assess blood inflammatory biomarkers (IL6, TNFa and IL1B) using enzyme-linked immunosorbent assay
Brain changes | pre- surgery (within five days before)
  Using non-invasive magnetic resonance imaging diffusion weighted (DW) pseudo-continuous arterial spin labeling (pCASL)
Brain changes II | Post-surgery (within two days post surgery)
  non-invasive magnetic resonance imaging diffusion weighted (DW) pseudo-continuous arterial spin labeling (pCASL)
Brain changes III | Post-surgery (within six months post surgery)
  Using non-invasive magnetic resonance imaging diffusion weighted (DW) pseudo-continuous arterial spin labeling (pCASL)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Kumar, Ph.D, Principal Investigator — rkumar@mednet.ucla.edu; Susana Vacas, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology & Perioperative Medicine, Los Angeles, California, United States